CLINICAL TRIAL: NCT07349706
Title: Randomized Controlled Pilot Trial of Inspiratory Muscle Strength Training (IMST) to Reduce Dementia Risk in Older Adults
Brief Title: IMST for Dementia Risk Reduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Julia Sheffler, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00006529
Record Dates: First submitted 2026-01-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Systolic Blood Pressure; Blood Pressure; Depression - Major Depressive Disorder; Anxiety; Sleep Quality; Physical Function; Cognitive Function
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High-Resistance (Experimental): Participants assigned to the high resistance arm will complete inspiratory muscle strength training (IMST) using a handheld respiratory training device set to 75% of their maximal inspiratory pressure (MIP). Participants will follow the IMST training regimen for the duration of the intervention period, 8-weeks, consisting of 30 breaths per day, completed in a minimum of 5 minutes.
  Interventions: Device: Inspiratory Muscle Strength Training
- Control Group - Low-Resistance (Sham Comparator): Participants assigned to the low-resistance arm will complete inspiratory muscle strength training (IMST) using a handheld respiratory training device set to 15% of their maximal inspiratory pressure (MIP). Participants will follow the IMST training regimen for the duration of the intervention period, 8-weeks, completing 30 inspiratory breaths per day, with each session lasting a minimum of 5 minutes.
  Interventions: Device: Inspiratory Muscle Strength Training

INTERVENTIONS:
Device: Inspiratory Muscle Strength Training — We will use POWERbreathe® Electronic IMST devices and manually set them to 75% or 15% of an individual's IPpeak, depending on their randomization, to the high-resistance IMST group or very low-resistance IMST (sham) group. All participants will complete 30 training breaths per day at home for 8 weeks.

SUMMARY:
Using a 2-arm, RCT approach, the primary goal of the study is to evaluate the feasibility and preliminary efficacy of Inspiratory Muscle Strength Training (IMST) as a non-pharmacologic intervention to reduce cardiovascular and cognitive risks in older adults. Next, we will examine secondary effects of IMST on mood, sleep quality, systemic inflammation, and physical/motor function. Finally, we will assess participant adherence and acceptability ratings of using an 8-week home-based IMST protocol in a diverse older adult sample.

DETAILED DESCRIPTION:
This is a 2-arm randomized pilot trial (N=30), including adults aged 60-80 years of age with cardiovascular risks for dements. Participants will complete assessments prior to beginning the study, each week during the intervention, and at the conclusion of the 8-week intervention. Participants in the experimental group will complete daily high-resistance IMST training (e.g., 75% maximal inspiratory pressure), and participants in the sham condition will complete IMST training at 15% maximal inspiratory pressure. We hypothesize the following: Hypothesis 1: Participants in the high-resistance IMST group will show greater reductions in systolic blood pressure and other vascular health indicators compared to those in the sham IMST group after 8 weeks.

Hypothesis 2: Participants in the high-resistance IMST group will demonstrate greater improvements in executive cognitive function than those in the sham group.

Hypothesis 3: IMST will lead to secondary improvements in mood (reduced depression and anxiety symptoms), better sleep quality (as measured by self-report and actigraphy), and improved physical function (e.g., grip strength, gait speed).

Hypothesis 4: The IMST protocol will be feasible and acceptable, with at least 80% adherence to prescribed training sessions over the 8-week period.

ELIGIBILITY:
Inclusion Criteria:

* Ages 60-80
* Converted telephone MoCA total score≥18
* Presence of at least one dementia risk factor (e.g., MCI or subjective cognitive decline, hypertension [SBP >130 mmHg or on medication], sedentary lifestyle [<150 min/week], family history of dementia or self-reported APOE ε4 carrier, or mild sleep-disordered breathing; CAIDE total score [>5]
* Capable of independently completing or requiring minimal assistance with inspiratory muscle strength training (IMST)
* Willing to adhere to the IMST protocol (approximately 5-10 minutes per day for 8 weeks)
* Optional inclusion of inspiratory muscle weakness (MIP <80 cmH₂O for men, <70 cmH₂O for women) will also be assessed.

Exclusion Criteria:

* tMoCA <18, or diagnosis of neurodegenerative illness at the discretion of principal investigator (except MCI)
* Current evidence of any major psychiatric disorder including psychosis (at the discretion of principal investigator), bipolar disorder, severe major depression (PHQ-9 > 20)
* Unstable cardiovascular or pulmonary disease
* Recent respiratory therapy or major medication changes
* Self-reported severe untreated or unstable obstructive sleep apnea (OSA)
* Recent start (within the past month) of CPAP or BiPAP, or recent use of inspiratory muscle training
* Lung and eardrum injuries
* Non-English speaking
* Participants with a pacemaker or other medical implants containing magnets or electronics will be noted and excluded from body composition analyses.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in systolic BP | Baseline, 8-weeks
  Participants will demonstrate a change in systolic blood pressure (mmHg), assessed as the average of two seated measurements obtained following two consecutive 5-minute rest periods, from baseline to post-intervention.
Change in executive cognitive functioning | Baseline, 8 weeks
  Participants will demonstrate a change in executive cognitive functioning, assessed using the Fluid Composite Score from the NIH Toolbox Cognition Battery. The Fluid Composite Score is derived from tasks assessing executive function, attention, working memory, episodic memory, and processing speed. Change in executive cognitive functioning will be evaluated as the difference in Fluid Composite Scores from baseline to post-intervention.

SECONDARY OUTCOMES:
Change from Baseline in Mood Symptoms (Depression and Anxiety) at 8 Weeks | Baseline, 8 weeks
  Participants will demonstrate a change in mood symptoms, assessed using the Patient Health Questionnaire-9 (PHQ-9) for depressive symptoms and the Geriatric Anxiety Scale (GAS) for anxiety symptoms. Change in mood symptoms will be evaluated as the difference in scores from baseline to 8 weeks, with higher scores indicating greater symptom severity.
Change from Baseline in Sleep Quality at 8 Weeks | Baseline, 8 weeks
  Participants will demonstrate a change in sleep quality, measured using the Pittsburgh Sleep Quality Index (PSQI) and objective sleep measures collected via actigraphy (Fitbit) devices provided to participants. Change in sleep quality will be evaluated as the difference in PSQI global scores, with higher scores indicating poorer sleep quality, and sleep metrics compiled from actigraphy data from baseline to 8 weeks.
Change from Baseline in Inflammatory Markers (CRP, IL-6, TNF-α) at 8 Weeks | Baseline, 8 weeks
  Participants will demonstrate a change in inflammatory markers, assessed from fasting blood samples. Serum concentrations of CRP, IL-6, and TNF-α will be measured using standardized laboratory analyses. Change in inflammatory markers will be evaluated from baseline to 8 weeks.
Change from Baseline in Physical Functioning at 8 Weeks | Baseline, 8 weeks
  Participants will demonstrate a change in physical functioning, assessed using grip strength, gait speed, and the sit-to-stand test. Change in physical functioning will be evaluated from baseline to 8 weeks based on performance across these standardized physical function measures. Higher grip strength, faster gait speed, and improved sit-to-stand performance indicate improved physical functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect the privacy and confidentiality of the participants.